CLINICAL TRIAL: NCT04056884
Title: A Randomized Controlled Group Intervention Trial for Siblings and Parents of Children With Chronic Illness (SIBS-RCT)
Brief Title: SIBS-Intervention for Siblings and Parents of Children With Chronic Illness
Acronym: SIBS-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Sykehuset Innlandet HF (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Krister W Fjermestad, Professor, University of Oslo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2018/2461
Record Dates: First submitted 2019-08-12; First posted 2019-08-14 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2024-04

CONDITIONS: Siblings of Children With Chronic Illness

STUDY DESIGN:
Intervention Model Description: Participants are randomized to intervention or 12-week waitlist. All participants who are randomized to waitlist will receive the intervention after waitlist.
Masking Description: N/A, not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SIBS intervention (Active Comparator): SIBS intervention is a 5-session group intervention for siblings and parents of children with chronic illness. Sessions 1-3 are delivered in one day, and sessions 4-5 are delivered in one day one week later.
  Interventions: Behavioral: SIBS intervention
- Waitlist (No Intervention): Waitlist is 12 week of no intervention/usual care

INTERVENTIONS:
Behavioral: SIBS intervention — SIBS is a manual-based group intervention for siblings and parents of children with chronic illness
  Arms: SIBS intervention

SUMMARY:
SIBS-RCT is a randomized controlled trial comparing the effect of a 5-session group intervention for siblings and parents of children with chronic illness to 12-week waitlist. Participants randomized to waitlist will receive the intervention after waitlist. The main outcome is sibling mental health, and secondary outcomes include family communication, sibling disorder knowledge, quality of life, and adaption. Outcomes will be examined at pre-, post, 3-, 6- and 12- month follow-up.

DETAILED DESCRIPTION:
Siblings' wellbeing is at risk when one's brother or sister has a neurodevelopmental disorder. Neurodevelopmental disorders are enduring somatic and/or mental conditions affecting the central nervous system, such as autism, intellectual disability, and cerebral palsy. The mechanisms behind the wellbeing risk for siblings are linked to siblings' lack of disorder knowledge, poor parental mental health due to extra care responsibilities, and impaired family communication. No evidence-based interventions to improve sibling wellbeing exist. To address this gap, we propose examining a group intervention for siblings and parents of children with neurodevelopmental disorders in a randomized controlled trial (SIBS-RCT). SIBS-RCT compares a 5-session manual-based sibling-parent group intervention delivered over two weeks, to 3-month "treatment as usual" waitlist. The planned sample is 288 siblings and 288 parents. Recruitment and intervention will take place in specialist and municipal health services. Inclusion criteria are being the sibling (aged 8-16 years) of a child (aged 0-18 years) who is diagnosed with neurodevelopmental disorder and who receives specialist or municipal health services. Participants will be randomized in blocks of 6 to intervention or waitlist. The primary outcome is sibling mental health. Secondary outcomes include quality of life, disorder knowledge, and family communication. Predictor measures include biological stress levels, parent mental health, disorder impairment, and group leader adherence to the SIBS-manual. Measures will be electronically rated by siblings, parents, and teachers at pre-intervention, post-intervention, and 3, 6, and 12 months follow-up. Main effects of the intervention will be measured as the mean mental health change difference between intervention and waitlist from pre-intervention to 3-month follow-up. We will also apply growth curve models to examine trajectories of outcomes from pre-intervention to 12-month follow-up. Expected outcomes include improved sibling wellbeing, improved health services for siblings and families of children with neurodevelopmental disorders, and better integration between municipal and specialist services.

ELIGIBILITY:
Inclusion Criteria:

1. Being the sibling of a child diagnosed with chronic illness who is aged 0 to 18 years and receives specialist and/or municipal health services.
2. One parent able to attend the intervention.

Exclusion Criteria:

1. Being enrolled as primary patients in specialist health services;
2. Chronic illness diagnosis.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 288 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Strengths and difficulties questionnaire (SDQ) | Pre to 12-months follow-up
  Sibling mental health, reported by siblings, parents, and main teacher

SECONDARY OUTCOMES:
Parent Child Communication Scale (PCCS) | Pre to 12-months follow-up
  Family communication, reported by siblings and parents
KINDL Fragebogen (KINDL) | Pre to 12-months follow-up
  Sibling quality of life, rated by siblings and parents
Sibling Knowledge Interview (SKI) | Pre to 12-months follow-up
  Sibling disorder knowledge based on brief interview
Negative Adjustment Scale (NAS) | Pre to 12-months follow-up
  Sibling adaption, reported by siblings

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norge, Norway

IPD SHARING:
Plan to Share IPD: No
The scientific advisory board for this trial involves researchers from multiple sites, and de-identified data will be shared although details are not set.

REFERENCES:
- [Derived] Schumann A, Vatne TM, Dalton L, Rapa E, Fjermestad KW. "It's like a car that doesn't like gasoline" - a qualitative study of siblings' understanding of anorexia nervosa in childhood: perspectives from siblings and parents. J Eat Disord. 2025 Oct 21;13(1):231. doi: 10.1186/s40337-025-01263-5. PMID 41121407
- [Derived] Kirchhofer SM, Fredriksen T, Orm S, Botta M, Zahl E, Cogo-Moreira H, Prentice CM, Vatne TM, Haukeland YB, Silverman WK, Fjermestad KW. Effectiveness of a group intervention to improve mental health in siblings of children with chronic disorders: a cluster randomized controlled trial. J Pediatr Psychol. 2025 Jun 1;50(6):443-453. doi: 10.1093/jpepsy/jsaf021. PMID 40146207
- [Derived] Fjermestad KW, Silverman WK, Vatne TM. Group intervention for siblings and parents of children with chronic disorders (SIBS-RCT): study protocol for a randomized controlled trial. Trials. 2020 Oct 14;21(1):851. doi: 10.1186/s13063-020-04781-6. PMID 33054825
- See also: Project website — http://www.sibs.no